CLINICAL TRIAL: NCT04076579
Title: Phase II Multi-Center Trial of Trabectedin in Combination With Olaparib in Advanced Unresectable or Metastatic Sarcoma
Brief Title: Trabectedin in Combination With Olaparib in Advanced Unresectable or Metastatic Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.132; HUM00161251 (Other: University of Michigan)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Sarcoma; Sarcoma Metastatic
MeSH Terms: conditions — Sarcoma | interventions — olaparib; Trabectedin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib + Trabectedin (Experimental): There are 2 cohorts. Both cohorts receive the same treatment:
  * Cohort 1: Leiomyosarcoma and liposarcoma
  * Cohort 2: Other bone or soft tissue sarcoma histologies
  Treatment consists of 21-day cycles for a maximum of 18 months.
  Interventions: Drug: Olaparib; Drug: Trabectedin

INTERVENTIONS:
Drug: Olaparib — Olaparib taken by mouth twice daily
Drug: Trabectedin — Trabectedin administered intravenously (IV) every 21 days

SUMMARY:
This phase II trial studies how well trabectedin and olaparib work in treating patients with sarcoma that cannot be removed by surgery or has spread to other places in the body. Drugs used in chemotherapy, such as trabectedin, work in different ways to stop the growth of tumor cells, either by killing cells, stopping them from dividing or stopping them from spreading. Olaparib may stop the growth of tumor cells by blocking pathways responsible for repairing damaged cells. Giving trabectedin and olaparib may shrink or stop the tumor from growing.

ELIGIBILITY:
Key Inclusion Criteria

* Age ≥ 16 years
* Advanced unresectable or metastatic sarcoma

  * Cohort 1: Leiomyosarcoma (LMS)/Liposarcoma (LPS)
  * Cohort 2: Other sarcoma histologies (excluding gastrointestinal stromal tumors)
* Received at least 1 prior standard chemotherapy. For cohort 1 patients, this must have included a prior anthracycline.
* Measurable disease by RECIST 1.1
* Adequate hematologic, renal, hepatic function
* Adequate creatine phosphokinase
* ECOG performance status ≤ 1
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (LLN)
* Women of childbearing potential and men must agree to use adequate contraception from signing informed consent to at least 6 months (females) and 5 months (men) after study drug treatment

Key Exclusion Criteria

* Prior therapy with PARP inhibitor, including olaparib
* Prior therapy with trabectedin
* Additional active malignancy or treatment for alternative cancer (excluding non-melanoma skin cancer) requiring treatment within the past two years
* Pregnant or breastfeeding women
* Known hypersensitivity to trabectedin or olaparib
* Other exclusions per protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Chugh, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1; Cohort 2: Both cohorts receive the same treatment:
  * Cohort 1: Leiomyosarcoma and liposarcoma
  * Cohort 2: Other bone or soft tissue sarcoma histologies Treatment consists of 21-day cycles for a maximum of 18 months. Olaparib: Olaparib taken by mouth twice daily Trabectedin: Trabectedin administered intravenously (IV) every 21 days
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 16 | 13
Completed | 12 | 9
Not Completed | 4 | 4
Not completed — Adverse Event | 2 | 0
Not completed — discontinued due to toxicity | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Patient was deemed ineligible before starting study treatment | 0 | 1
Not completed — Noncompliance | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1; Cohort 2: Both cohorts received the same treatment:
  * Cohort 1: Leiomyosarcoma and liposarcoma
  * Cohort 2: Other bone or soft tissue sarcoma histologies Treatment consists of 21-day cycles for a maximum of 18 months. Olaparib: Olaparib taken by mouth twice daily Trabectedin: Trabectedin administered intravenously (IV) every 21 days
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Percentage of participants with complete or partial response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, within each cohort.
Time Frame: Up to 2 years
Population: one patient in cohort 2 was not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 12
Participants | 0 | 2

2. Secondary Outcome: Progression Free Survival
Description: Defined as the duration of time from start of treatment to time of progression. Calculated by the Kaplan-Meier method with errors according to Peto, within each cohort. Median and 6-month PFS will be estimated along with their 95% confidence intervals.
Time Frame: At 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 12
months | 4.1 [3.3 to NA] — not reportable per biostatistician. The "NA" values appear because the upper confidence limit for the median could not be estimated. The upper confidence limit requires the upper confidence bound of the survival curve to fall below 50 percent. If it remains above 50 percent throughout follow-up, the upper limit cannot be estimated and will be reported as "NA" or "NE." This is what happened here. | 3.8 [2.2 to NA] — not reportable per biostatistician. The "NA" values appear because the upper confidence limit for the median could not be estimated. The upper confidence limit requires the upper confidence bound of the survival curve to fall below 50 percent. If it remains above 50 percent throughout follow-up, the upper limit cannot be estimated and will be reported as "NA" or "NE." This is what happened here.

3. Secondary Outcome: Progression Free Survival
Description: Defined as the duration of time from start of treatment to time of progression. Calculated by the Kaplan-Meier method with errors according to Peto, within each cohort. reported as survival probability estimates
Time Frame: At 1 year after enrollment
Measure: Number; unit: percentage of patients
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 12
percentage of patients | 8.9 | 20.2

4. Secondary Outcome: Overall Survival
Description: Calculated by the Kaplan-Meier method with errors according to Peto, within each cohort. Median, 1- and 2-year OS probability estimates will be estimated along with their 95% confidence intervals.
Time Frame: At 2 years after enrollment
Measure: Number (95% Confidence Interval); unit: probability estimates
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 12
probability estimates
  1 year post enrollment | 0.52 [0.28 to 0.94] | 0.48 [0.24 to 0.94]
  2 year post enrollment | 0 [0 to 0] | 0.12 [0.02 to 0.74]

5. Secondary Outcome: Incidence of Adverse Events
Description: The frequency and rates of adverse events occurring in at least 5% of participants and rates of grade 3-5 adverse events will be tabulated by system organ class and preferred term using Common Terminology Criteria of Adverse Events (CTCAE), within each cohort.
Time Frame: Up to 30 days after end of treatment, and average of 4.5 months
Measure: Number; unit: number of events
Groups:
- Cohort 1; Cohort 2: Both cohorts receive the same treatment:
  Cohort 1: Leiomyosarcoma and liposarcoma Cohort 2: Other bone or soft tissue sarcoma histologies Treatment consists of 21-day cycles for a maximum of 18 months. Olaparib: Olaparib taken by mouth twice daily Trabectedin: Trabectedin administered intravenously (IV) every 21 days
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 14
number of events
  Acute Kidney Injury- Grade 3 | 0 | 1
  Alanine aminotransferase increased- Grade 3 | 1 | 3
  Anemia- Grade 3 | 5 | 1
  Aspartate aminotransferase increased - Grade 3 | 1 | 1
  Blood bilirubin increased- Grade 3 | 1 | 0
  Bronchopulmonary hemorrhage - Grade 3 | 0 | 1
  Ejection fraction decreased- Grade 4 | 0 | 1
  Fatigue- Grade 3 | 2 | 0
  Fever- Grade 3 | 1 | 0
  Hypokalemia- Grade 3 | 0 | 1
  Lung Infection- Grade 3 | 0 | 1
  Lymphocyte count decreased- Grade 3 | 0 | 1
  Myalgia- Grade 3 | 1 | 0
  Neutrophil count decreased- Grade 3 | 31 | 8
  Neutrophil count decreased- Grade 4 | 11 | 9
  Platelet count decreased- Grade 3 | 8 | 1
  Platelet count decreased- Grade 4 | 3 | 0
  Sepsis- Grade 3 | 1 | 0
  Sinus tachycardia- Grade 3 | 0 | 1
  White blood cell decreased- Grade 3 | 11 | 1
  White blood cell decreased- Grade 4 | 4 | 1

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 3 year period.
Description: Adverse Events and All-Cause Mortality will be evaluated with secondary endpoints as data is still being collected.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 10/16 | 5/13
Serious Adverse Events (participants affected / at risk) | 2/16 | 4/13
Other Adverse Events (participants affected / at risk) | 16/16 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=16) | Cohort 2 (N=13)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=16) | Cohort 2 (N=13)
Abdominal pain (General disorders) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (13) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3)
Allergic reaction (General disorders) | 1 (1) | 0 (0)
Anemia (Investigations) | 11 (28) | 6 (15)
Anorexia (Psychiatric disorders) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 3 (6)
Back pain (General disorders) | 2 (2) | 0 (0)
Blood bilirubin increased (Hepatobiliary disorders) | 2 (3) | 0 (0)
Bruising (General disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Creatinine increased (Investigations) | 6 (9) | 1 (5)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (2)
Dysgeusia (General disorders) | 2 (2) | 0 (0)
Dyspepsia (General disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Fatigue (General disorders) | 14 (19) | 4 (6)
Fever (General disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhoids (General disorders) | 1 (1) | 0 (0)
Hiccups (General disorders) | 1 (1) | 0 (0)
Hypocalcemia (Investigations) | 1 (1) | 1 (2)
Hypokalemia (Investigations) | 1 (1) | 1 (2)
Mucositis oral (General disorders) | 2 (2) | 0 (0)
Myalgia (General disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (15) | 4 (5)
Neutrophil count decreased (Investigations) | 13 (56) | 7 (25)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 9 (27) | 6 (17)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Sore throat (General disorders) | 1 (1) | 0 (0)
Thrush (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2)
Weight loss (General disorders) | 2 (3) | 1 (1)
White blood cell decreased (Investigations) | 7 (23) | 3 (8)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1)
Hyperglycemia (Investigations) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Investigations) | 0 (0) | 1 (3)
Hyponatremia (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2)
Memory impairment (General disorders) | 0 (0) | 1 (1)
Nasal congestion (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04076579/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT04076579/ICF_001.pdf